CLINICAL TRIAL: NCT07062445
Title: Prospective Clinical Registry of Acute Treatment and Long-term Assessment of Children Meningitis
Acronym: ATLAS-II
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: ATLAS-II
Record Dates: First submitted 2025-05-29; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Meningitis; Bacterial Infections; Viral Meningitis; Fungal Meningitis
Keywords: meningitis; bacterial; virus; corticosteroids; antibiotics; fungal
MeSH Terms: conditions — Meningitis; Bacterial Infections; Meningitis, Viral; Meningitis, Fungal; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Biospecimen Retention: Samples Without DNA — serum and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicenter, observational clinical registry of pediatric patients with acute infectious meningitis across approximately 20 public and private hospitals in Brazil. The study will include children under 18 years of age with suspected acute infectious meningitis. Data will be collected during hospitalization and post-discharge to evaluate clinical management, treatment and short and long-term outcomes. The study aims to generate real-world evidence on current practices and outcomes to support improvements in national care protocols.

DETAILED DESCRIPTION:
This is a middle-income real-world prospective clinical registry study. Clinical and laboratory data will be collected during hospitalization and follow-up visits will be performed at 28, 90 and 180 days after inclusion in the study.

Data collection will include empirical antibiotic therapy timing and type, time from hospital admission to antibiotic's first dose, corticosteroid therapy initiation, vaccination status per the Brazilian National Immunization Program (PNI), neurological sequelae and access to specialized rehabilitation services post-discharge.

Primary outcomes will be all-cause mortality, length of hospital stay, rate of re-hospitalization and sensorineural hearing loss incidence.

Secondary outcomes will be etiology-specific mortality, functional outcomes (PCPC-BR and pediatric FSS - Brazilian version), guideline-based therapies by etiology, neurological sequelae incidence stratified by etiology (e.g., motor deficits, cerebrovascular complications) , serious adverse events and access to rehabilitation.

Findings will be used to inform public health system and pediatric clinical care in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Fever (axillary temperature ≥37.8°C) followed by two or more of the following symptoms*: severe headache, vomiting, altered consciousness (confusion, drowsiness, or irritability), photophobia (increased sensitivity to light), presence of seizures OR
* Fever accompanied by at least one meningeal irritation sign, such as neck stiffness, Kernig's sign, or Brudzinski's sign OR
* Sudden onset of fever and appearance of petechial skin rash or hemorrhagic suffusions

  * In children younger than two years, in addition to the presentations listed above, consider fever with any of the following: irritability, persistent crying, somnolence, or bulging fontanelle.

Exclusion Criteria:

* Refusal to provide consent for study participation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population, <17 years old, suspect of acute meningitis infection
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mortality, re-hospitalization, length of hospital stay and sensory hearing loss | Day 28
  The primary outcome is a composite endpoint and for that a hierarchical statistical analysis of the components will be applied, considering their clinical importance and the temporal relevance between events (mortality will take precedence over the other components: incidence of all-cause re-hospitalization, length of initial hospital stay -measured in days and incidence of sensory hearing loss). The statistical methodology will include the use of the hierarchical Win Ratio and/or equivalent approaches.

SECONDARY OUTCOMES:
Patients with guideline-directed therapy | Day 180
  Proportion of patients receiving empirical and targeted therapies according to national meningitis management guidelines
Mortality in six months | Day 180
  Incidence of all-cause mortality
Rate of re-hospitalization | Day 180
  Incidence of all-cause re-hospitalization
Invasive ventilatory support | Day 28
  Incidence of invasive ventilatory support
Access to specialized rehabilitation services post-discharge | Day 28, day 90 and day 180
  Proportion of patients receiving specialized rehabilitation care
Length of hospitalization by etiology | Day 180
  Length of hospitalization (in days), stratified by infectious etiology
Re-hospitalization rate by etiology | Day 180
  Rate of unplanned re-hospitalization stratified by etiology
Neurological sequelae by etiology | Day 180
  Incidence of neurological sequelae stratified by etiology
Post-discharge functional neurological decline | Day 28 and day 180
  Neurological Functional Status will be assessed using Brazilian version of the Functional Status Scale (FSS-BR):
  * No disability: FSS= 6
  * Mild disability: FSS= 7-9
  * Moderate disability: FSS= 10-15
  * Severe disability: FSS= 16-21
  * Very severe disability: FSS>21
Cerebral Performance Post-Meningitis | Day 28 and day 180
  Cerebral Performance Post-Meningitis will be assessed using PCPC-BR (Pediatric Cerebral Performance Category - Brazilian version).
  For the purpose of this analysis, cases with a score of 6 (brain death) will be excluded here, as they will be accounted separately in the mortality outcome.
  * No disability: PCPC= 1
  * Mild disability: PCPC= 2
  * Moderate disability: PCPC= 3
  * Severe disability: PCPC= 4
  * Very severe disability: PCPC=5
Adverse Events | Day 28
  Incidence of adverse events
Adverse outcomes by etiology | Day 180
  Incidence of adverse outcomes by etiology

CONTACTS AND LOCATIONS:
Overall Officials: Henrique A Fonseca, Study Chair — Hospital Israelita Albert Einstein; Anna M Gomes, Principal Investigator — Hospital Israelita Albert Einstein

IPD SHARING:
Plan to Share IPD: No